CLINICAL TRIAL: NCT00690976
Title: Proyecto SOL: A Risk Reduction Intervention for Hispanic MSM
Brief Title: Proyecto SOL: A Risk Reduction Intervention for Hispanic Men Who Have Sex With Men (MSM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Nova Southeastern University (Other); University of Miami (Other); DePaul University (Other)
Responsible Party: Isa fernandez, Prinicpal Investigator, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-5123
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV risk behavior; Unprotected sex; men who have sex with men; gay; Latino; Unsafe Sex
MeSH Terms: conditions — HIV Infections; Unsafe Sex; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.Group Intervention (Experimental): A group-based intervention consisting of 4 sessions lasting approximately 90 minutes each. Using a variety of pedagogical and interactive approaches, facilitators will introduce new concepts and skills.
  Interventions: Behavioral: Proyecto SOL
- 2. HCT (Active Comparator): Offer of HIV counseling and testing
  Interventions: Behavioral: HCT

INTERVENTIONS:
Behavioral: Proyecto SOL — Group intervention
  Arms: 1.Group Intervention
Behavioral: HCT — Offer of HIV counseling and testing
  Arms: 2. HCT

SUMMARY:
The purpose of this project is to determine the acceptability, feasibility, and the preliminary efficacy of an HIV prevention behavioral intervention (Proyecto SOL) to reduce behaviors associated with HIV acquisition among Hispanic men who have sex with men (HMSM). The primary goal of the intervention is to motivate and assist participants in forming and carrying out a "Safer Options for Life" plan, thereby reducing their risk of HIV acquisition or transmission.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Hispanic or Latino;
* be between 18 and 49 years of age;
* be a resident of South Florida (Miami-Dade, Broward or Palm Beach counties) and not planning to move out of the area for the next 9 months;
* self-identify as male;
* have had at least one episode of unprotected anal sex with a man in the preceding 3 months;
* have had 2 or more male sex partners in the preceding 3 months;
* be HIV negative or of unknown serostatus;
* speak English and/or Spanish;
* provide informed consent.

Exclusion Criteria:

* have previously participated in any Phase of this study;
* self-identify as transgender;
* not being a resident of South Florida.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Unprotected sex | three months

CONTACTS AND LOCATIONS:
Overall Officials: Isa Fernandez, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- NOVA Southeastern University, Fort Lauderdale, Florida, United States